CLINICAL TRIAL: NCT02573610
Title: A Randomized, Double-masked, Parallel Group Study of DE-108 Ophthalmic Solution in Patients Who Are Scheduled for Cataract Surgery (Levofloxacin 0.5% Ophthalmic Solution as a Comparator) - Phase III, Confirmatory Study of Perioperative Bacteria Eradication -
Brief Title: Study of DE-108 Ophthalmic Solution in Patients Who Are Scheduled for Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DE-108
Record Dates: First submitted 2015-10-07; First posted 2015-10-12 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Cataract Surgery
MeSH Terms: interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DE-108 (Experimental): High concentration / Antibacterial Ophthalmic Solution
  Interventions: Drug: DE-108
- Levofloxacin 0.5% (Active Comparator): Low concentration / Antibacterial Ophthalmic Solution
  Interventions: Drug: Levofloxacin 0.5%

INTERVENTIONS:
Drug: DE-108 — Subjects will be assigned to receive DE-108 ophthalmic solution to be administrated one drop a time 3 times daily for 3 days prior and for 14 days following cataract surgery.
  Other Names: Levofloxacin
  Arms: DE-108
Drug: Levofloxacin 0.5% — Subjects will be assigned to receive Levofloxacin 0.5% ophthalmic solution to be administrated one drop a time 3 times daily for 3 days prior and for 14 days following cataract surgery.
  Arms: Levofloxacin 0.5%

SUMMARY:
The purpose of this study is to evaluate superior efficacy of DE-108 ophthalmic solution to that of Levofloxacin 0.5% ophthalmic solution as well as safety of the former used for perioperative bacteria eradication in patients who are scheduled for cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Those who are scheduled for cataract surgery

Exclusion Criteria:

* Those who with suspected ocular infections based on clinical findings in the study eye.
* Those who have any eye disease other than cataract which requires treatment in the target eye.
* Those who have a history of allergy to the drugs to be used during the clinical study (such as fluoroquinolones, topical anesthetics and povidon iodine)
* Those who need to wear contact lenses during the study period

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Change in the percentage of positive bacteriological test results (from Day -3 to Day 0) | 3 days (Day -3 to Day0)

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Kyungpook National University Hospital, Kyungpook
  - Asan Medical Center, Seoul
  - Kim's eye Hospital, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul Saint Marry's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul